CLINICAL TRIAL: NCT04874649
Title: Effects of Balloon Blowing Breathing Exercise on Respiratory Muscle Strength and Symptoms in School-age Children With Asthma.
Brief Title: Balloon Blowing Breathing Exercise in School-age Children With Asthma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EX PHYSIO SPSC 1
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Asthma in Children
Keywords: Balloon blowing breathing; respiratory muscle strength; school-age children with asthma; Sustained maximal inspiration (SMI) breathing; Asthma symptoms
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Thirty school-age children with asthma aged 7 - 12 years old who were admitted at the outpatient examination room, Phramongkutklao Hospital, divided into 2 groups. The first group was 15 individuals trained with sustained maximal inspiration (SMI) breathing exercise while the second group was 15 individuals training with balloon-blowing breathing exercise. Participants were required to complete breathing exercise 5 times per week for 8 weeks. Physiological characteristics data and pulmonary function variables were comparatively analyzed before and after training. The dependent variables between pre-test and post-test were analyzed by a paired t-test. Independent t-test was used to compare the variables between groups. Differences were considered to be significant at p < .05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon-blowing breathing (Experimental): 1. Start by measuring the vital capacity using a balloon to determine. The width of the balloon diameter for each blow and used the value to make a balloon size control device to give to the sample group and parents to use it for home training.
  2. Participant sit on a chair. Inhale fully through their nose and hold for a full 3 second inhalation, then exhale through their mouth into the balloon fully. By having the balloon inflate until their touch the balloon size control device and hold the exhalation period for 1 second, cover the balloon immediately with your fingers count as 1 breath cycle, then replace the balloon immediately. Do this for 3 consecutive rounds, counted as 1 set, in each training, do a total of 3 sets, rest between sets for 1 minute, which takes about 15 minutes, 5 times per week for 8 weeks
  Interventions: Other: Balloon-blowing breathing
- Sustained maximal inspiration breathing (Experimental): Participants sitting in a chair, back and head close to the wall. Inhale through their nose fully and hold for 3 seconds for a full breath, then slowly exhale through their mouth and hold for 1 second of exhalation, counted as 1 breathing cycle.Do this 3 times in a row for 1 set. Practice each time doing a total of 3 sets, with 1 minute rest between sets. Participants were required to complete breathing exercise 5 times per week for 8 weeks.
  Interventions: Other: Sustained maximal inspiration breathing

INTERVENTIONS:
Other: Balloon-blowing breathing — Participant sit on a chair. Inhale fully through their nose and hold for a full 3 second inhalation, then exhale through their mouth into the balloon fully. By having the balloon inflate until their touch the balloon size control device and hold the exhalation period for 1 second, cover the balloon immediately with your fingers count as 1 breath cycle, then replace the balloon immediately. Do this for 3 consecutive rounds, counted as 1 set, in each training, do a total of 3 sets, rest between sets for 1 minute, which takes about 15 minutes, 5 times per week for 8 weeks
  Arms: Balloon-blowing breathing
Other: Sustained maximal inspiration breathing — Participant sit on a chair. Inhale through their nose fully and hold for 3 seconds for a full breath, Do this for 3 consecutive rounds, counted as 1 set, in each training, do a total of 3 sets, rest between sets for 1 minute, which takes about 15 minutes, 5 times per week for 8 weeks
  Arms: Sustained maximal inspiration breathing

SUMMARY:
This study were to investigate the effects of balloon blowing breathing exercise on respiratory muscle strength and asthma symptoms in school-age children with asthma.

DETAILED DESCRIPTION:
Thirty school-age children with asthma aged 7 - 12 years old who were admitted at the outpatient examination room, Phramongkutklao Hospital, divided into 2 groups. The first group was 15 individuals trained with sustained maximal inspiration (SMI) breathing exercise while the second group was 15 individuals training with balloon-blowing breathing exercise. Participants were required to complete breathing exercise 5 times per week for 8 weeks. Five breathing exercises were taken for 8 weeks before and after the experiment. Physiological characteristics data, pulmonary function, respiratory muscle strength, and asthma symptoms variables were comparatively analyzed before and after training. The mean values of variables before and after the experiment of each group were analyzed using paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* has been diagnosed with asthma for at least 6 months. The severity rating is not higher than level 2, (Forced expiratory volume in one second; FEV1 is at least 80%)
* No history of diabetes, heart disease, and musculoskeletal disease
* Did not participate in exercise training for more than 20 minutes 3 times a week or more in the 6 months prior to the start of data collection.

Exclusion Criteria:

* Patient with a history of exercise-induced asthma.
* Recurrent of acute exacerbation
* Cannot participate at least 80% of training program (≤ 32 sessions of 40 sessions)
* Unwilling to continue practicing

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength change | Change from Baseline respiratory muscle strength at 8 weeks.
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds.
Asthma control change | Change from Baseline Asthma control at 8 weeks.
  Asthma control was measured by Childhood Asthma Control Test (C - ACT) questionnaire. The range of C-ACT scores is 0 to 27 (27 = totally controlled, 20-26 = well controlled, <26 = insufficiently controlled)

SECONDARY OUTCOMES:
Force Vital Capacity (FVC) change | Change from Baseline Force Vital Capacity at 8 weeks.
  FVC is the total volume of air that can be exhaled during a maximal forced expiration effort. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FVC is measured in liters.
Forced expiratory volume in 1 second (FEV1) change | Change from Baseline Forced expiratory volume in 1 second at 8 weeks.
  FEV1 is the volume of air exhaled in the first second under force after a maximal inhalation. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEV1 was showed in liters.
The ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) change | Change from Baseline The ratio of forced expiratory volume in 1 second to forced vital capacity at 8 weeks.
  It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC). The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEV1/FVC was showed in percentage.
Peak Expiratory Flow (PEF) change | Change from Baseline Peak Expiratory Flow at 8 weeks.
  PEF is the amount and rate of air that can be forcefully breathed out of the lungs. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. PEF is measured in liters/seconds.
Forced Expiratory Flow from 25% to 75% of vital capacity (FEF25-75%) change | Change from Baseline Forced Expiratory Flow from 25% to 75% of vital capacity (FEF25-75%) at 8 weeks.
  FEF25-75% is the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEF25-75% is forced expiratory flow over the middle one half of the FVC; the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled. FEF25-75% is measured in liters/seconds.
Maximal Voluntary Ventilation (MVV) change | Change from Baseline Maximum Voluntary Ventilation at 8 weeks.
  The participants were asked to inhale and exhale quickly and forcefully for 10 seconds. Maximal Voluntary Ventilation (MVV) were measured in liters/minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Background] Chauhan, N., & Gunjal, S. (2018). Effect of Balloon Blowing Exercise on Peak Expiratory Flow Rate in Modified Radical Mastectomy. International Journal of Health Sciences & Research, 8(10).
- [Background] Collins JE, Gill TK, Chittleborough CR, Martin AJ, Taylor AW, Winefield H. Mental, emotional, and social problems among school children with asthma. J Asthma. 2008 Aug;45(6):489-93. doi: 10.1080/02770900802074802. PMID 18612902
- [Background] Das, S. M., Nayak, G. R., & Pradhan, R. (2018). Effect of Balloon Therapy vs. Bubble Therapy on LRTI among 3-12 Years Children. International Journal of Health Sciences & Research, 8(1), 144-147.
- [Background] Gomieiro LT, Nascimento A, Tanno LK, Agondi R, Kalil J, Giavina-Bianchi P. Respiratory exercise program for elderly individuals with asthma. Clinics (Sao Paulo). 2011;66(7):1163-9. doi: 10.1590/s1807-59322011000700007. PMID 21876968
- [Background] Grammatopoulou EP, Skordilis EK, Stavrou N, Myrianthefs P, Karteroliotis K, Baltopoulos G, Koutsouki D. The effect of physiotherapy-based breathing retraining on asthma control. J Asthma. 2011 Aug;48(6):593-601. doi: 10.3109/02770903.2011.587583. Epub 2011 Jun 13. PMID 21668321
- [Background] Jun HJ, Kim KJ, Nam KW, Kim CH. Effects of breathing exercises on lung capacity and muscle activities of elderly smokers. J Phys Ther Sci. 2016 Jun;28(6):1681-5. doi: 10.1589/jpts.28.1681. Epub 2016 Jun 28. PMID 27390394
- [Background] Kang JI, Jeong DK, Choi H. The effects of breathing exercise types on respiratory muscle activity and body function in patients with mild chronic obstructive pulmonary disease. J Phys Ther Sci. 2016 Jan;28(2):500-5. doi: 10.1589/jpts.28.500. Epub 2016 Feb 29. PMID 27064889
- [Background] Lima EV, Lima WL, Nobre A, dos Santos AM, Brito LM, Costa Mdo R. Inspiratory muscle training and respiratory exercises in children with asthma. J Bras Pneumol. 2008 Aug;34(8):552-8. doi: 10.1590/s1806-37132008000800003. English, Portuguese. PMID 18797738
- [Background] Marcelino AM, da Cunha DA, da Cunha RA, da Silva HJ. Respiratory muscle strength in asthmatic children. Int Arch Otorhinolaryngol. 2012 Oct;16(4):492-6. doi: 10.7162/S1809-97772012000400010. PMID 25991978